CLINICAL TRIAL: NCT05403528
Title: Technological Timescales: Identifying the Impact of Digital Media on the Mechanisms of Word Learning
Brief Title: Technology/Digital Media Use and Children's Word Learning Development
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: original clinical trials form had error, but cannot be deleted at this stage
Sponsor: Oklahoma State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sarah Kucker, Assistant Professor, Oklahoma State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AS-18-155; R15HD101841 (NIH)
Record Dates: First submitted 2022-05-23; First posted 2022-06-03 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of for conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3D-3D (No Intervention): All items presented in 3D form
- 3D-2D (Experimental): Initial items in 3D, retention and generalization in 2D
  Interventions: Behavioral: Modality - 3D-2D
- 2D-3D (Experimental): Initial items in 2D, retention and generalization in 3D
  Interventions: Behavioral: Modality - 2D-3D
- 2D-2D (Experimental): All items in 2D
  Interventions: Behavioral: Modality - 2D-2D

INTERVENTIONS:
Behavioral: Modality - 3D-2D — Modality in which items will be presented (via tablet/digital media or as real object). 3D items initially and retention/generalization as 2D
  Other Names: digital media modality
  Arms: 3D-2D
Behavioral: Modality - 2D-3D — Modality in which items will be presented (via tablet/digital media or as real object). 2D items initially and retention/generalization as 3D
  Other Names: digital media modality
  Arms: 2D-3D
Behavioral: Modality - 2D-2D — Modality in which items will be presented (via tablet/digital media or as real object). 2D items initially and retention/generalization as 2D
  Other Names: digital media modality
  Arms: 2D-2D

SUMMARY:
The goal of this work is to address increasing concerns about young children's digital media exposure and language outcomes by testing how the times course of word learning unfolds in digital environments and the cascading impact of digital media on vocabulary outcomes. The findings will have important implications for understanding when and where optimal word learning from media can occur.

DETAILED DESCRIPTION:
The goal of the current proposal is to identify how digital media alters the mechanisms of word learning and subsequently impacts the lexical foundation on which a child's vocabulary is built. Specifically, the proposal aims to identify the impact of digital media on 1) the processes underlying real-time word learning, and 2) the processes of language generalization and vocabulary growth. Specific Aim 1 will use a novel word learning task to test children's ability to map and retain new words within and between digital media (2D images on a tablet) and real world objects (3D objects). Specific Aim 2 will probe children's novel label generalization abilities within and between 2D and 3D modalities using a novel noun generalization task. Further, individual differences in a child's prior technology experience will be measured and used to predict overall vocabulary as well as performance within and between each task.

ELIGIBILITY:
Inclusion Criteria:

* between 17-30 months old

Exclusion Criteria:

* diagnosed developmental delay or disorder
* exposure to more than 25% of another language

Ages: 17 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Accuracy on selecting the target item on referent selection | 1 minute
  Children's choices on each trial of the task will be measured. Correct responses are those to the target (prompted) item - for referent selection, this is the item asked for in the prompt (e.g. shoe, dog)
Accuracy on selecting the target item on retention | 5 minutes
  Children's choices on each trial of the task will be measured. Correct responses are those to the target (prompted) item - for retention, this is the item asked for in the prompt.
Accuracy on selecting the target item on novel noun generalization task | 1 minute
  Children's choices on each trial of the task will be measured. Correct responses are those to the target (prompted) item - for generalization this will be considered as the shape-matching item (and not choosing a color or material match)

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Studies proposed will be registered under the Open Science Framework (OSF) and resulting findings shared with the academic community through open science initiatives, including OSF and the sharing of videos (when permission is granted) on Databrary.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After completion of the project and for the duration allowed by the IRB.
Access Criteria: Databrary authorized user